CLINICAL TRIAL: NCT05211505
Title: Prospective, Open-label Trial Investigating the Efficacy and Tolerability of WO 2707, a MoistCream Cremolum, in Postmenopausal Women Suffering From Symptoms of Vaginal Dryness
Brief Title: Investigation of Efficacy and Tolerability of WO 2707, a MoistCream Cremolum, in Postmenopausal Women Suffering From Symptoms of Vaginal Dryness
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dr. August Wolff GmbH & Co. KG Arzneimittel (Industry)
Collaborators: proDERM GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VFCrC-01/2021
Record Dates: First submitted 2022-01-13; First posted 2022-01-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Vaginal Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WO 2707 (Experimental): Formulation containing WO 2707 for intravaginal application
  Interventions: Device: WO 2707

INTERVENTIONS:
Device: WO 2707 — Intravaginal application once daily for 1 week, then twice per week until visit 3 (day 38).

SUMMARY:
The objective of the clinical investigation is to evaluate the efficacy and tolerability of WO 2707, a MoistCream Cremolum, with respect to the application in postmenopausal women with symptoms of vaginal dryness.

ELIGIBILITY:
Inclusion Criteria:

1. Post-menopausal women with the subjective symptomatology of vulvovaginal atrophy with a sum score (0-16) of the parameters dryness, itching, burning and pain unrelated to sexual intercourse of at least 3 AND a score of at least "2" (moderate) for the parameter dryness at screening and visit 1 (day 1)

   * Thereof at least for 48 included patients: sexual activity with dyspareunia
   * Thereof at least 32 included sexually active patients with at least moderate (score of "2") dyspareunia
2. Natural cessation of last menstruation more than 12 months before screening OR bilateral oophorectomy with or without hysterectomy more than 3 months before screening
3. Signed written informed consent before participation in the clinical investigation

Exclusion Criteria:

1. Vaginal inflammation which is not caused by vulvovaginal atrophy
2. Non-healed vaginal surgery
3. Systemic hormonal replacement therapy (tablets, patches, injections, dermal products), or phytohormonal therapy or use of SERMs (selective estrogen receptor modulators) within 3 months before visit 1 (day 1) and / or during the conduct of this clinical investigation
4. Local hormonal therapy (vagina/vulva) within 3 months before Screening (also when used for the brightening/pretreatment of cytological smears)
5. Any use of products (including lubricants), other than the investigational medicinal device, applied intravaginally or on the vulva during the clinical investigation (except usual cleansing products)
6. Systemic corticosteroids within 21 days before visit 1 (day 1) and during the conduct of this clinical investigation (corticoid asthma sprays are allowed)
7. Use of antibiotics, antiseptics or antimycotics with expected or suspected systemic or vaginal/vulvar bioavailability within 21 days before visit 1 (day 1) and / or during this clinical investigation
8. Known hypersensitivity against any of the ingredients of the investigational medical device
9. Employees of the investigation sites who are directly involved in this clinical investigation or employees of the sponsor's company

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participant eligibility based on self-representation of gender identity.
Enrollment: 79 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2022-03-24 (Actual); Study Completion 2022-03-24 (Actual)

PRIMARY OUTCOMES:
Change of TSS (Total severity score) for subjective symptoms of atrophy | From baseline to visit 3 (day 38)
  The severity of each of the subjective symptoms dryness, itching, burning and pain unrelated to sexual intercourse will be assessed according to the following scale: 0=none, 1=mild, 2=moderate, 3=severe, 4=very severe
  The total severity score will be calculated as the sum score of the subjective symptoms resulting in a minimum score of 0 (best) and a maximal score of 16 (worst).

SECONDARY OUTCOMES:
Change of TSS (Total severity score) for subjective symptoms of atrophy | From baseline to visit 2 (day 8), visit 2 (day 8) to visit 3 (day 38) and visit 3 (day 38) to visit 4 (day 44)
  The severity of each of the subjective symptoms dryness, itching, burning and pain unrelated to sexual intercourse will be assessed according to the following scale: 0=none, 1=mild, 2=moderate, 3=severe, 4=very severe
  The total severity score will be calculated as the sum score of the subjective symptoms resulting in a minimum score of 0 (best) and a maximal score of 16 (worst).
Change of severity scoring for each of the subjective symptoms (dryness, itching, burning and pain unrelated to sexual intercourse) | From baseline to visit 2 (day 8) and visit 3 (day 38), visit 2 (day 8) to visit 3 (day 38) and visit 3 (day 38) to visit 4 (day 44)
  The severity of each of the subjective symptoms dryness, itching, burning and pain unrelated to sexual intercourse will be assessed according to the following scale: 0=none, 1=mild, 2=moderate, 3=severe, 4=very severe
Change of each DIVA domain score (A - D) and change of total DIVA score (excluding questions 12 to 15) | From baseline to visit 3 (day 38)
  The DIVA questionnaire addresses the impact of vaginal symptoms such as vaginal dryness, soreness, irritation and itching on the day-to-day life regarding the patient's activities, relationships, and feelings by any of these symptoms (Huang, 2015; Gabes, 2021).
Change of each DIVA domain score (A - D) and change of total DIVA score in the subgroup of sexually active women with dyspareunia | From baseline to visit 3 (day 38)
  The DIVA questionnaire addresses the impact of vaginal symptoms such as vaginal dryness, soreness, irritation and itching on the day-to-day life regarding the patient's activities, relationships, and feelings by any of these symptoms (Huang, 2015; Gabes, 2021).
Change of each single parameter and of sum score over objective assessment of VHI | From baseline to visit 3 (day 38)
  The objective status of the vagina will be assessed by the Investigator according to the Vaginal Health Index (Bachmann, 1995). Each of the five criteria - elasticity, fluid secretion, pH, epithelial mucosa and moisture - will be graded from 1 (worst) to 5 (best) and will then be summed up, so that the minimum score will be 5 (worst) and the maximum score will be 25 (best)
Change of vaginal pH | From baseline to visit 3 (day 38)
Patient questionnaire | Day 3, visit 3 (day 38), visit 4 (day 44)
Change of severity scoring for dyspareunia for the subgroup of sexually active women with dyspareunia | From baseline to visit 2 (day 8) and visit 3 (day 38), visit 2 (day 8) to visit 3 (day 38) and visit 3 (day 38) to visit 4 (day 44)
  Severity scoring for Dyspareunia will be assessed by the patients according to the following scale: 0=none,1=mild, 2=moderate, 3=severe, 4=very severe
Change of impairment of daily life due to dyspareunia (VAS) for the subgroup of sexually active women with dyspareunia | From baseline to visit 2 (day 8) and visit 3 (day 38), visit 2 (day 8) to visit 3 (day 38) and visit 3 (day 38) to visit 4 (day 44)
  Impairment of daily life due to dyspareunia will be assessed using a 10 cm visual analogue scale (VAS) ranging from 0 (no impairment) to 10 (very pronounced impairment).
Global judgement of efficacy by the investigator | On visit 3 (day 38)
  The global judgement of efficacy will be assessed according to the following scale: 1=very good, 2=good, 3=moderate, 4=poor
Global judgement of efficacy by the patient | On visit 3 (day 38)
  The global judgement of efficacy will be assessed according to the following scale: 1=very good,2=good, 3=moderate, 4=poor
Global judgement of tolerability by the investigator | On visit 3 (day 38)
  The global judgement of tolerability will be assessed according to the following scale: 1=very good, 2=good, 3=moderate, 4=poor
Global judgement of tolerability by the patient | On visit 3 (day 38)
  The global judgement of tolerability will be assessed according to the following scale: 1=very good, 2=good, 3=moderate,4=poor
Participants with premature trial termination due to adverse device effects, adverse events, concomitant medication | From baseline to visit 4 (day 44)

CONTACTS AND LOCATIONS:
Overall Officials: Kirstin Deuble-Bente, MD, Principal Investigator — proderm GmbH, Germany
Locations (1):
- proderm GmbH, Schenefeld, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eichler S, Panz M, Harder A, Masur C, Hauser M, Wiesche ESZ. An effective non-hormonal option with high tolerability for mild to moderate symptoms of vaginal dryness associated with menopause. Maturitas. 2024 Jul;185:107978. doi: 10.1016/j.maturitas.2024.107978. Epub 2024 Mar 29. PMID 38583316
- [Derived] Gabes M, Donhauser T, Harder A, Masur C, Apfelbacher CJ. Psychometric evaluation of the German Day-to-Day Impact of Vaginal Aging questionnaire using data from two intervention studies. Menopause. 2023 May 1;30(5):551-555. doi: 10.1097/GME.0000000000002161. Epub 2023 Feb 14. PMID 36787527